CLINICAL TRIAL: NCT05966753
Title: Observational Study on the Management, and Progression of Patients With Diabetic Macula Edema (DME)
Brief Title: Describing Patient With DME, Their Patient Journey and Disease Progression
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1485-0016
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diabetic macula edema (DME): Patients diagnosed with diabetic macula edema (DME) in at least one eye, at least 18 years old, with information on laterality and registered in the Vestrum health database between January 2015 and May 2023.

SUMMARY:
This study aims to characterize patients with diabetic macular edema (DME), their progression, the treatment received and associate the functional and physiological outcomes related to the treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients ≥18 years, with a DME diagnosis in at least one eye, included in the Vestrum database identified during the study period (January 2015 to April 2023)

Exclusion Criteria:

Patients without the information of laterality will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is based on the patients attending a retinal specialist, included in the Vestrum Retinal specialist database. The study population will include adult patients with a DME diagnosis in at least one eye.
Sampling Method: Non-Probability Sample
Enrollment: 221004 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity | From January 2015 to April 2023
Progression to DME in the fellow eye | From January 2015 to April 2023
Initial treatment of DME | From January 2015 to April 2023
Central retinal thickness (CRT) | From January 2015 to April 2023

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas HQ, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com